CLINICAL TRIAL: NCT01645449
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-way Crossover Oral BE Study of Atorvastatin Ca 80 mg Tablets of Dr. Reddy's and Lipitor 80 mg Tablets of Pfizer in Healthy Adult, Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Atorvastatin Calcium Tablets, 80 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-VIN-095
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Atorvastatin calcium; crossover
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin Calcium Tablets, 80 mg (Experimental): Atorvastatin Calcium Tablets, 80 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Atorvastatin Calcium Tablets, 80 mg
- Lipitor 80 mg Tablets (Active Comparator): Lipitor 80 mg Tablets of Pfizer Ireland Pharmaceuticals
  Interventions: Drug: Atorvastatin Calcium Tablets, 80 mg

INTERVENTIONS:
Drug: Atorvastatin Calcium Tablets, 80 mg — Atorvastatin Calcium Tablets, 80 of Dr. Reddy's Laboratories Limited
  Other Names: Lipitor 80 mg Tablets

SUMMARY:
The purpose of this study is to compare and evaluate the single-dose oral bioavailability and to monitor the safety of subjects.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-way crossover oral bioequivalence' study of Atorvastatin Calcium 80 mg Tablets of Dr. Reddy's and Lipitor 80 mg Tablets of Pfizer Ireland Pharmaceuticals in healthy adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 - 55 (including) years old.
2. Subjects' weight within normal range according to normal values for Body Mass Index (1 8.0 to 30.0 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within clinically acceptable range.
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. systolic blood pressure between 90 mmHg to 145 mmHg (age 18 to 45 years) or 90 mmHg to 160 mmHg (above 45 years). Diastolic blood pressure between 50 mrnHg to 90 rnmHg. Pulse rate between 45 bpm and 100 bpm.
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and morphine).
7. Subjects having negative alcohol breath test.
8. Women who are of childbearing potential must be using acceptable methods of birth control for 4 weeks prior to, during and 4 weeks after the last dose of trial medication and should be informed of the potential risks associated with becoming pregnant while enrolled within a clinical research trial. Accepted forms of contraception are: i.e. implants, injectables, hormonal intrauterine device, combined oral contraceptives, sexual abstinence and vasectomised sexual partner throughout the trial. Female volunteers who are post-menopausal, hysterectomised or surgically sterile may be enrolled.
9. Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

The subjects were excluded from the study, if they met any of the following criteria:

1. Hypersensitivity to the test, or reference drug, or all other used ingredients, or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological,neurological or psychiatric disease or disorder.
3. Individual or farniliy case medical history of any myopathy.
4. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month before first dosing in Period 1.
5. Medical history of muscular toxic reactions during treatment with statins of fibrates.
6. Use of any prescribed or OTC medication or herbal supplements within 14 days or within 5 times the half-life of the respective active substance (whatever is longer), before first dosing in Period 1 (excluding contraceptives on women).
7. History or presence of significant alcoholism or drug abuse in the past one year. Alcoholism is defined as consumption of more than 50g of ethanol per day (12.5 cL glass of 10° [l0%]] wine = 12 g; 4 cL of aperitif, 42° [42 %] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g.
8. History or presence of significant smoking (more than 10 cigarettes/day).
9. History or presence of asthma, urticaria or other significant allergic reactions.
10. History or presence of significant gastric andlor duodenal ulceration.
11. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
12. History or presence of cancer.
13. Difficulty with donating blood.
14. Difficulty in swallowing solids like tablets or capsules.
15. Major illness during 3 months before first dosing in Period 1.
16. Participation in a drug research study within the past 1 month before first dosing in Period 1.
17. Donation of blood in the past 2 months before first dosing in Period 1.
18. Consumption of grapefruit juice, xanthine-containing products or alcohol for within 48 hours prior to dosing.
19. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
20. History or presence of significant easy bruising or bleeding.
21. History or presence of significant recent trauma.
22. Pregnancy or breast-feeding (for female subjects).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose at 0.00 hour and post-dose at 0.167, 0.333, 0.50, 0.667, 0.833, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.50, 2.75, 3.00, 3.50, 4.00,6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00 and 72.00 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Margarete Muller, Principal Investigator — Nuvisan Pharma Services GmbH & Co. KG
Locations (1):
- Nuvisan Pharma Services GmbH & Co. KG, Neu-Ulm, Germany